CLINICAL TRIAL: NCT01138267
Title: Impact of Pharmacogenomics on Antiretroviral Drugs (Atazanavir and Efavirenz) Concentration and Treatment Response in HIV-infected Adults Study-team
Brief Title: Pharmacogenomic of Atazanavir/Efavirenz (ATV/EFV)
Status: Completed | Type: Observational
Sponsor: The HIV Netherlands Australia Thailand Research Collaboration (Other)
Collaborators: Chulalongkorn University (Other); Kirby Institute (Other Government); Radboud University Medical Center (Other); SEARCH Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: HIV-NAT103
Record Dates: First submitted 2010-06-04; First posted 2010-06-07 (Estimated); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: HIV Infections
Keywords: pharmacogenomics; ATV; EFV; pharmacogenomics of ATV and EFV
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Patients are divided into 4 groups based on whether they need to redraw their blood.
  1. have adequate samples stored and do not need additional blood draws.
  2. have EFV or ATV blood concentrations samples stored but do not have samples for genotyping. Need extra 5-ml sample.
  3. have samples stored but the samples cannot be used to test for EFV or ATV blood concentrations because the time of drug intake and blood drawn are unknown. Need to redraw 5-ml sample.
  4. have never had both drug concentration and genotyping done. Need to give 10 ml of blood sample to perform both tests.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Objectives:

* To evaluate the impact of genetic polymorphism on ARV drug levels
* To evaluate the effect of genetic polymorphism/drug levels on long term immunologic and virologic response
* To correlate the genetic polymorphism/drug levels on antiretroviral toxicities

The long-term objective of this research plan is to characterize impact of pharmacogenomics to HIV drug concentration, toxicities, and response to antiretroviral therapy among HIV-infected adults. A comprehensive understanding of the impact of pharmacogenomics to HIV infection and HIV medication will lead to the development of appropriate intervention such as dose reduction strategies in patients with particular gene(s) correlated with higher drug levels. The dose reduction strategy will decrease long term drug toxicity and cost saving for Thais and Asian Ethnicities.

DETAILED DESCRIPTION:
The overall goal of this study is to characterize role of pharmacogenomic on ARV drug (atazanavir, and efavirenz) levels, its toxicities, and its long term efficacy among HIV-infected adults in Thailand. The specific aims are (1) to evaluate the impact of genetic polymorphism on ARV drug levels (2) to evaluate the effect of genetic polymorphism/ drug levels on long term immunologic and virologic response (3) to correlate the genetic polymorphism/drug levels on antiretroviral toxicities. The proposed study will be analysed in stored samples of the well-established cohort of long-term follow-up study for HIV-infected patients participated in HIV-NAT study protocols, the HIV-NAT006 study. This cohort provide us unique opportunity to study impact of pharmacogenomics on long term treatment response and long term drug toxicities since this cohort was started in 1996. Furthermore, the important factors include ARV regimen, drug toxicities, PBMC, immunological and virological parameters have been collected every 6 months basis in HIV-NAT006 study.

A comprehensive understanding of the impact of pharmacogenomics to HIV infection and HIV medication will lead to development of appropriate intervention, particularly, dose reduction strategy in patient with particular gene correlated with greater drug levels. The dose reduction strategy will decrease long term drug toxicity and cost saving for Thai and Asian Ethnicity.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for pharmacogenomic of ATV:

1. On low-dose ATV/r at the time blood samples are collected for ATV drug levels
2. Age > 18 years of age or older with HIV-1 infection
3. Provided consent form

Inclusion criteria for pharmacogenomic of EFV:

* On EFV at the time blood samples are collected for EFV levels
* Age > 18 years of age or older with HIV-1 infection
* Patients who were on EFV but later switched to another ARV regimen due to toxicity of EFV and have stored sample at time of taking EFV
* Provided consent form

Exclusion Criteria:

Exclusion criteria for both ATV and EFV

1. Inability to understand the nature and extent of the study and the procedures required.
2. Contramedication such as rifampin, proton pump inhibitor (for ATV), etc
3. Pregnancy during blood drawn for EFV or ATV drug levels
4. Known renal insufficiency or cirrhosis during blood drawn for EFV or ATV drug levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected participants previously or currently enrolled in any HIV-NAT trials since 1996
Sampling Method: Non-Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Frequency of MDR1-3435 allele variants,MDR1-2677 allele variants,UGT1A1 allele variants, frequency of CYP 2B6 variants in efavirenz treatment and compare candidate gene and treatment response of ATV/r or EFV | 2 years

SECONDARY OUTCOMES:
Compare drug conc. of UGT1A1 variant with bilirubin, drug conc. & treatment resp. of ATV/r or EFV, drug conc.for WT, drug conc.for 2B6 variant with EFV toxicity & drug discontinuation, drug conc.or 2B6 variant with long term efficacy & EFV resistance | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, Principal Investigator — Chulalongkorn University
Locations (1):
- HIV-NAT Thai Red Cross AIDS Research Center, Bangkok, Thailand

REFERENCES:
- [Derived] Chaivichacharn P, Avihingsanon A, Manosuthi W, Ubolyam S, Tongkobpetch S, Shotelersuk V, Punyawudho B. Dosage Optimization of Efavirenz Based on a Population Pharmacokinetic-Pharmacogenetic Model of HIV-infected Patients in Thailand. Clin Ther. 2020 Jul;42(7):1234-1245. doi: 10.1016/j.clinthera.2020.04.013. Epub 2020 May 22. PMID 32451120
- See also: HIV Netherland Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org